CLINICAL TRIAL: NCT06568978
Title: Evaluation of Disease Severity, Respiratory Muscle Strength, Respiratory Functions, Functionality, and Quality of Life in Patients With Upper Limb Lymphedema
Brief Title: Evaluation of Respiratory Parameters in Patients With Upper Limb Lymphedema
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Okan University (Other)
Responsible Party: Principal Investigator, Gamze Aydin, Researcher, PhD, Istanbul University - Cerrahpasa
Other Study IDs: IstanbulOU
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Lymphedema of Upper Limb
Keywords: Lymphedema; upper limb; quality of life; respiratory function test
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: patients with upper limb lymphedema
  Interventions: Other: Assessments of respiratory parameters
- Group 2: healthy individuals
  Interventions: Other: Assessments of respiratory parameters

INTERVENTIONS:
Other: Assessments of respiratory parameters — respiratory muscle strength, respiratory function test

SUMMARY:
The aim of our study is to assess disease severity, respiratory muscle strength, respiratory functions, pectoralis minor muscle shortening, functionality, and quality of life (QoL) in patients with upper limb lymphedema (ULL), and to compare these findings with healthy controls.The disease severity was assessed using the Stillwell classification system; respiratory muscle strength was measured through maximum inspiratory and expiratory intraoral pressures (MIP, MEP, respectively); respiratory functions were evaluated with a spirometer; pectoralis minor muscle shortening was measured with a tape measure; functionality was assessed using the Disabilities of the Arm, Shoulder and Hand (DASH); and QoL was evaluated with the Lymphedema Quality of Life Questionnaire - Arm (LYMQOL-Arm).

DETAILED DESCRIPTION:
The study had a cross-sectional observational study design. The participants were divided into two groups, patients with ULL in Group 1; the healthy individuals were included in Group 2. All assessments for both groups were performed by two different physiotherapists.

ELIGIBILITY:
Inclusion Criteria:

* aged 25-65 years with secondary, unilateral upper limb lymphedema in Phase 2 of the protection stage,
* wearing compression garments,
* who have not received manual lymph drainage (MLD) therapy in the last 3 months
* along with healthy controls of a similar age who volunteered to participate.

Exclusion Criteria:

* being in Phase 1 of lymphedema treatment (the edema-reducing phase),
* being classified as NYHA Class III and/or IV according to the New York Heart Association classification system,
* having a chronic respiratory disease,
* presence of active infection (such as lymphangitis or cellulitis), or undergoing radiotherapy/chemotherapy due to breast cancer.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: aged 25-65 years with secondary, unilateral upper limb lymphedema patients and healthy controls
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
MIP and MEP value | 9 months
  assessments include maximal inspiratory intraoral pressure (MIP) and expiratory intraoral pressure (MEP).
FVC | 9 months
  FVC is used for forced vital capacity which measure by spirometer
pectoralis minor muscle length | 9 months
  pectoralis minor muscle length is used for pectoralis muscle shortness
DASH questionnaire | 9 months
  Disabilities of the Arm, Shoulder and Hand (DASH) is used for upper extremity functions. Questionnaire score ranged between 0-100. A higher total score indicates decreased functionality.
LYMQOL-Arm questionnaire | 9 months
  Lymphedema Quality of Life Questionnaire - Arm is used for assess disease related quality of life.The high scores are indicative of poorer QoL. Questionnaire score ranged between 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Aydın, PhD, Principal Investigator — Okan University
Locations (1):
- Gamze Aydın, Tuzla, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided